CLINICAL TRIAL: NCT06803264
Title: Effectiveness of Activity Oriented Therapy and Traditional Therapy in Cervical Discopathic Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40/KBL/OIL/2020
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2023-06

CONDITIONS: Neck Pain Chronic; Depression Disorders; Forward Head Posture; Anxiety Disorders
Keywords: N.A.P. therapy, breathing exercises, neuroplasticity, forward head posture, chronic neck pain, psychosomatic diseases.
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N.A.P. therapy group (Experimental): Activity Oriented therapy (N.A.P.) is based on the assumption that motor activity affects the plasticity of the brain and it stimulates a positive change in its cortical representation. The therapist use motor teaching techniques, postural control exercises and improving respiratory functions. Breathing exercises are used to reduce nervous system stimulation, activating the parasympathetic system and relaxing the body and mind. Additionally, diaphragm exercises affect the stabilization of the spine muscles.
  Interventions: Other: Activity Oriented therapy (N.A.P.)
- Traditional therapy group (Active Comparator): In Poland, traditional treatment of neck pain includes physical treatments (e.g. cryotherapy or TENS) and exercises to strengthen and improve the range of muscles in the shoulder girdle and neck. Research shows that these interventions provide good benefits in the treatment of neck pain immediately after therapy, but there is often a lack of information about how this change is maintained over time. Considering the psychological aspect of chronic pain, such actions may not be sufficient to effectively cure the problem.
  Interventions: Other: Traditional therapy

INTERVENTIONS:
Other: Activity Oriented therapy (N.A.P.) — The following six exercises were used, each of which was performed 10 times. Their progression was introduced by changing positions, individually adjusted to the patient's capabilities.
  1. Eccentric infrahyoid muscle work during breathing activity and phonation of the "l"sound.
  2. Reciprocal innervation of suboccipital muscles in gaze activity.
  3. Stimulation of the diaphragm in the activity of breathing and phonation.
  4. Repeated eccentric activity of the sternocleidomastoid (SCM) muscles during body transfer activity.
  5. Repeated eccentric activity of scalene muscles in blanket pulling activity.
  6. Eccentric work of suboccipital muscles in the activity of biting a snack.
  Arms: N.A.P. therapy group
Other: Traditional therapy — Traditional therapy included:
  1. Isometric work of the neck muscles.
  2. Self-assisted active exercises for the shoulder girdle muscles.
  3. Active exercises in relief for the muscles of the shoulder girdle performed in the sitting position in the transverse plane.
  4. TENS current treatment performed in the cervical spine and shoulder girdle in the forward lying position.
  5. The local cryotherapy treatment with carbon dioxide.
  Arms: Traditional therapy group

SUMMARY:
Title: Effectiveness of Activity Oriented Therapy and Traditional Therapy in Cervical Discopathic Pain Syndrome

Procedures: You will be asked to complete a form containing questions characterizing the study group and several questionnaires before starting treatment, such as: NDI, CESD-R, STAI and the NRS scale. A photo of the head and shoulder area will also be taken in a front and side standing position. After completing the two-week treatment, you will be asked again to complete questionnaires and pose for photos. You will be informed about a follow-up visit 3 months after the end of therapy, during which you will be asked for the last time to complete questionnaires and pose for a photo.

Benefits: There are no direct benefits to you other than participating in a therapy more commonly used for cervical pain syndromes and the opportunity to discuss your experience with neck pain with a specialist. The information we obtain will help scientists better understand the problem of treating neck pain.

Risk: There are no physical risks to you while conducting this research. All information obtained from you will be anonymous. Your name and image will not be used in this study or reports.

Confidentiality: All research records will be confidential and appropriately secured. Records will only be published with your consent or by court order or as required by law. Any publication resulting from this research will not use identifying information, such as your name or likeness.

Freedom to opt out: Participation in the study is completely voluntary and free of charge. You may withdraw from this study at any time without any consequences.

DETAILED DESCRIPTION:
The purpose of the study was to evaluate the effectiveness of the Activity Oriented Therapy (N.A.P. therapy) and traditional therapy during disc-related neck pain in terms of pain intensity, disability, Forward Head Posture (FHP), anxiety as a condition and level of depression. Patients were qualified based on a medical examination. Respondents were randomly divided into two groups.

The therapies were performed by experienced physiotherapists in cooperation with a psychologist. Treatment in both groups included 10 therapy sessions held daily from Monday to Friday over a two-week period.

ELIGIBILITY:
Inclusion Criteria:

* qualifying: non-traumatic, disc-like, chronic (symptoms lasting more than 3 months) cervical pain of mechanical origin, localized in the cervical region with the possibility of radiation to the upper edge of the scapula and head (without root symptoms and neurological disorders), classified as syndrome No. 1 according to the Quebec Task Force (QTF) Classification, and a condition not requiring surgery.

Exclusion Criteria:

* comorbid advanced neurological, rheumatic, urological, psychiatric diseases, and unsystematic participation in in therapy.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NRS) | Before therapy, after two weeks of treatment and after 3 months of follow-up
  The Numerical Rating Scale (NRS), which contains 11 levels of pain intensity, where 0 means no pain and 10 means maximum pain
The Neck Disability Index (NDI) | Before therapy, after two weeks of treatment and after 3 months of follow-up
  The Neck Disability Index (NDI) questionnaire, which examines the level of disability from NP. A patient can score between 0 and 50 points. A score between 1-4 points indicates no disability, 5-14 points mild disability, 15-24 points moderate disability, 25-34 points severe disability, and above 35 points total disability.
The photographic method to assess Forward Head Posture (FHP) | Before therapy, after two weeks of treatment and after 3 months of follow-up
  The photographic method to assess FHP. Based on photographs of the shoulder area and head taken in the forward and lateral standing positions, two angles were measured using the computer program GIMP (version 2.10.34). The camera was placed on a tripod at a distance of 150 cm from the patient. Cranio Vertebral Angle (CVA) was measured in the sagittal plane, while Frontal Head Tilt angle (FHT) was measured in the frontal plane. A higher score for CVA and a lower score for FHT indicate improvement in FHP. The reliability of the described procedure is rated as high. In the author's study, images were taken with a SONY DSC-W810B camera.
The State-Trait Anxiety Inventory (STAI) | Before therapy, after two weeks of treatment and after 3 months of follow-up
  The State-Trait Anxiety Inventory (STAI), which examines the level of anxiety understood as a transient and situationally conditioned state of the individual and anxiety as a relatively stable personality trait. The STAI consists of two subscales, but only the scale for measuring anxiety-state (X-1) was used in this study. Each subscale can be scored from 20 to 80. High values indicate higher levels of anxiety.
The Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) | Before therapy, after two weeks of treatment and after 3 months of follow-up
  The Center for Epidemiologic Studies Depression Scale-Revised (CESD-R). This is a self-report scale that examines levels of depression. It consists of 20 statements relating to mood and behavior observed over the past two weeks. The lowest score is 0 and the highest score is 80. The higher the scores, the higher the level of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Clinic "Azory", Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The article includes data such as age, gender and duration of symptoms.

REFERENCES:
- [Background] Szczygiel E, Fudacz N, Golec J, Golec E. The impact of the position of the head on the functioning of the human body: a systematic review. Int J Occup Med Environ Health. 2020 Sep 17;33(5):559-568. doi: 10.13075/ijomeh.1896.01585. Epub 2020 Jul 23. PMID 32713947
- [Background] Jerath R, Beveridge C. Respiratory Rhythm, Autonomic Modulation, and the Spectrum of Emotions: The Future of Emotion Recognition and Modulation. Front Psychol. 2020 Aug 14;11:1980. doi: 10.3389/fpsyg.2020.01980. eCollection 2020. PMID 32922338
- [Background] Maric V, Ramanathan D, Mishra J. Respiratory regulation & interactions with neuro-cognitive circuitry. Neurosci Biobehav Rev. 2020 May;112:95-106. doi: 10.1016/j.neubiorev.2020.02.001. Epub 2020 Feb 3. PMID 32027875
- [Background] Nitayarak H, Charntaraviroj P. Effects of scapular stabilization exercises on posture and muscle imbalances in women with upper crossed syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2021;34(6):1031-1040. doi: 10.3233/BMR-200088. PMID 34151819
- [Background] Schuch FB, Vancampfort D, Richards J, Rosenbaum S, Ward PB, Stubbs B. Exercise as a treatment for depression: A meta-analysis adjusting for publication bias. J Psychiatr Res. 2016 Jun;77:42-51. doi: 10.1016/j.jpsychires.2016.02.023. Epub 2016 Mar 4. PMID 26978184
- [Background] Cohen SP, Hooten WM. Advances in the diagnosis and management of neck pain. BMJ. 2017 Aug 14;358:j3221. doi: 10.1136/bmj.j3221. PMID 28807894
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Elman I, Borsook D. Common Brain Mechanisms of Chronic Pain and Addiction. Neuron. 2016 Jan 6;89(1):11-36. doi: 10.1016/j.neuron.2015.11.027. PMID 26748087